CLINICAL TRIAL: NCT03429088
Title: Exercise Promotion in Primary Care: Pilot Study
Brief Title: Exercise Promotion in Primary Care
Acronym: EPPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Deborah R. Young, Research Scientist III, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KPSC IRB#10106
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2018-02

CONDITIONS: Physical Activity; PreDiabetes; Diabetes
MeSH Terms: conditions — Motor Activity; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone counseling (Experimental): Participants were provided with approximately 7 telephone-based motivational interviewing over a 24-week period to increase their physical activity.
  Interventions: Behavioral: Motivational interviewing telephone counseling
- Usual care (No Intervention): Participants in the usual care arm received a packet of places near their home in which they could engage in physical activity if they chose.

INTERVENTIONS:
Behavioral: Motivational interviewing telephone counseling
  Arms: Telephone counseling

SUMMARY:
The investigators conducted a pilot study to determine if telephone counseling, in a health care setting that routinely assesses physical activity of its members, is a feasible approach to improve physical activity among patients with diabetes and prediabetes. The investigators built on an existing innovation at Kaiser Permanente, in which physical activity is assessed at every outpatient visit. The primary aims were to (1) pilot study elements, including database identification of patients; recruitment, training and engagement of health care providers; patient recruitment; data collection procedures; and a 24-week intervention, and (2) to assess feasibility and obtain feedback from key stakeholders on the approach.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes or diabetes not prescribed insulin
* less than 30 min of physical activity per week
* cleared to increase physical activity by primary care provider

Exclusion Criteria:

* health condition that may limit unsupervised physical activity
* height and weight that were combined and resulted in a BMI > 40 kg/m2
* disabling rheumatoid or osteoarthritis
* ongoing treatment for cancer
* unstable coronary heart disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of identifying and recruiting sufficient number of participants into a telephone-based physical activity intervention. | The intervention lasted 24 weeks.
  Participants who met eligibility criteria and who were scheduled for an outpatient visit with their primary care provider were invited to participate in the study. Feasibility was assessed by the investigators' ability to recruit 60 participants into the pilot trial.

SECONDARY OUTCOMES:
Moderate to Vigorous Physical Activity | Assessments were made a baseline and approximately 24 weeks after baseline assessments.
  Participants were mailed an Actigraph model 7185 accelerometer and asked to wear it over their right hip for 7 consecutive days and return the monitor through the mail. Data were analyzed to assess daily moderate to vigorous physical activity using the Freedson cutpoints.
Motivation for Physical Activity | Participants completed the survey at baseline and approximately 24 weeks after baseline assessments.
  The 30-item Motivation for Physical Activities Measure was used to measure motivation for physical activity. The scale has 5 factors: interest/enjoyment, competence, appearance, fitness, and social motivations. A mean score for each factor was determined for each participant.
Physical Activity Self-Regulation | Participants completed the survey at baseline and approximately 24 weeks after baseline.
  This is a 16-item scale with the following factors: external regulation, introjected regulation, identified regulation, and intrinsic regulation. A Relative Autonomy Index is formed from the factors, with the higher scores indicating greater autonomy toward physical activity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young DR, Nguyen MK, Yamamoto A, Pomichowski M, Cornejo M, Paz S, Coleman KJ, Sallis RE, Fortmann SP. Telephone-based motivational interviewing versus usual care in primary care to increase physical activity: a randomized pilot study. Pilot Feasibility Stud. 2019 Jan 15;5:6. doi: 10.1186/s40814-019-0390-0. eCollection 2019. PMID 30675373